CLINICAL TRIAL: NCT04279002
Title: Association of Psycho-social Traits for the Benefit of a First Respiratory Rehabilitation Course - Exploratory Study.
Acronym: RESPIRSO
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19/RESPIRSO; 2019-A02774-53 (Other: IdRCB)
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Rehabilitation; Pulmonary Rehabilitation
Keywords: Personality traits; Anxiety; Depression; Social support
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Respiratory rehabilitation course: Patients who has completed at least one respiratory rehabilitation course at the Espace du Souffle (Tours France) within the 5 years prior to inclusion
  Interventions: Other: Brief 15-question questionnaire

INTERVENTIONS:
Other: Brief 15-question questionnaire — Questionnaire is mailed retrospectively to the respiratory rehabilitation program and aimed at targeting 17 psycho-social traits. Response time is estimated at 10 minutes

SUMMARY:
Respiratory Rehabilitation (RR) is based on a comprehensive multidisciplinary program of personalized and tailored care for patients with chronic respiratory diseases.

The effectiveness of RR in improving quality of life and exercise capacity has long been demonstrated in patients with chronic obstructive pulmonary disease (COPD). More recently, its interest has been highlighted in other chronic respiratory pathologies: asthma, interstitial pathologies, cancer, restrictive pathologies or pulmonary arterial hypertension. Although the efficacy of RR has been well demonstrated on the scale of a patient population, the benefits derived on an individual scale remain unpredictable and variable from one individual to another, without knowing the major determinants of this benefit.

Empirically, RR professionals suspect an association between some psychosocial characteristics and the importance of the benefit derived by patients from RR programmes. Individual personality traits and their relationship to health status, integration into a group, interaction with other group members, and the existence of anxiety or depressive symptoms may be determinants of RR benefit. These psychosocial determinants could also play a central role in the patients' adherence to the long-term rehabilitation process.

The hypothesis being tested is that there is an association between personality traits, anxiety, depressive symptoms, social support, and the benefit of an initial course of RR and the subsequent continuation of maintenance practices.

DETAILED DESCRIPTION:
Respiratory Rehabilitation (RR) is based on a comprehensive multidisciplinary program of personalized and tailored care for patients with chronic respiratory diseases. Carried out in small groups of patients, it offers effort re-training combined with therapeutic education and psychological and social care. It aims at the long-term change of life habits.

The effectiveness of RR in improving quality of life and exercise capacity has long been demonstrated in patients with chronic obstructive pulmonary disease (COPD). More recently, its interest has been highlighted in other chronic respiratory pathologies: asthma, interstitial pathologies, cancer, restrictive pathologies or pulmonary arterial hypertension. Although the efficacy of RR has been well demonstrated on the scale of a patient population, the benefits derived on an individual scale remain unpredictable and variable from one individual to another, without knowing the major determinants of this benefit.

Empirically, RR professionals suspect an association between some psychosocial characteristics and the importance of the benefit derived by patients from RR programmes. Individual personality traits and their relationship to health status, integration into a group, interaction with other group members, and the existence of anxiety or depressive symptoms may be determinants of RR benefit. These psychosocial determinants could also play a central role in the patients' adherence to the long-term rehabilitation process.

The hypothesis being tested is that there is an association between personality traits, anxiety, depressive symptoms, social support, and the benefit of an initial course of RR and the subsequent continuation of maintenance practices.

Main objective n°1: to describe the distribution of 17 psychosocial traits of interest in patients who had a major benefit from the initial RR stage (defined by a decrease ≥7 points of Saint George's Respiratory Questionnaire (SGRQ) compared to patients who did not have a major benefit (defined by a decrease <7 points of the SGRQ).

The 17 traits describe the following:

1. Personality traits
2. Existence of anxiety or depressive symptoms
3. Self-assessment of health status and the degree of control that the subject feels he or she has over the disease.
4. Felt social support
5. Interpersonal dimensions
6. General satisfaction of the subject

Secondary Objective 1 :

Describe the distribution of the 17 psychosocial traits of interest in patients who have implemented maintenance practices for at least one year after the 1st RR course (defined by paramedical care or participation in activities offered by a patient association or declaration of the maintenance of supervised physical activity), compared to patients who have not pursued such an activity or for whom this data is not available.

Secondary objective n°2: Describe the correlations between 17 psychosocial traits of interest and the variation of the following variables between the initial and final assessment of the first RR stage: SGRQ, VQ11 quality of life score, Modified Medical Research Council (mMRC) dyspnea scale, 6-minute walking distance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Completion of at least one respiratory rehabilitation course at the Espace du Souffle (Tours France) within the 5 years prior to inclusion.
* Participation Agreement (no opposition confirmed with the return of the questionnaire)

Exclusion Criteria:

* Protected adults (guardianship or trusteeship)
* Patient having expressed a refusal of contact for scientific purposes at the Espace du Souffle (Tours France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a chronic respiratory pathology and having carried out a respiratory rehabilitation program in the 5 years prior to inclusion at the Espace du Souffle in Tours (France).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Distribution of 17 psychosocial traits of interest in patients who had a major benefit from the initial Respiratory Rehabilitation program | At the inclusion
  Patients who had a major benefit from the initial Respiratory Rehabilitation program is defined by a decrease ≥7 points of the SGRQ
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.

SECONDARY OUTCOMES:
Distribution of the 17 psychosocial traits of interest in patients who have implemented maintenance practices for at least one year after the 1st Respiratory Rehabilitation program | At the inclusion
  Maintenance practices being defined by paramedical care or participation in activities offered by a patient association or declaration of continued supervised physical activity), compared to patients who have not pursued such an activity or for whom this data is not available.
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.
Assess correlations between between 17 psychosocial traits of interest and the variation of the SGRQ between the initial and final assessment of the first Respiratory Rehabilitation program | At the inclusion
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.
Assess correlations between between 17 psychosocial traits of interest and the variation of the VQ11 quality of life score between the initial and final assessment of the first Respiratory Rehabilitation program | initial and final assessment of the first Respiratory Rehabilitation program
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.
Assess correlations between between 17 psychosocial traits of interest and the variation of the mMRC dyspnea scale between the initial and final assessment of the first Respiratory Rehabilitation program | At the inclusion
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.
Assess correlations between between 17 psychosocial traits of interest and the variation of the 6-minute walking distance between the initial and final assessment of the first Respiratory Rehabilitation program | At the inclusion
  The 17 psycho-social traits are assessed using a short 15-item questionnaire mailed retrospectively to the Respiratory Rehabilitation Program.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent PLANTIER, MD-PhD, Study Director — University Hospital, Tours
Locations (1):
- Espace du Souffle, Tours, France